CLINICAL TRIAL: NCT00114374
Title: SSRI Administration to Reduce Acute Stress Disorder Symptoms and Prevent Depression and Posttraumatic Stress Disorder in Physical Trauma Victims in the Medical Setting
Brief Title: SSRI Administration to Reduce Acute Stress Disorder Symptoms and Prevent Depression and PTSD in Physical Trauma Victims
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Naomi M. Simon, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2004-P-001633
Record Dates: First submitted 2005-06-14; First posted 2005-06-15 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety Disorder
Keywords: Acute Stress Disorder; Posttraumatic Stress Disorder; Escitalopram; Double-Blind
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Traumatic, Acute; Stress Disorders, Post-Traumatic | interventions — Escitalopram

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
The purpose of this study is to examine the efficacy of escitalopram compared to placebo in reducing Acute Stress Disorder (ASD) symptoms and in preventing the emergence of Post-Traumatic Stress Disorder (PTSD) in patients with medical trauma who are at risk for the development of PTSD based on the presence of ASD symptoms.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a relatively common, distressing and disabling condition that may occur after trauma related events including injury. The emergence of Acute Stress Disorder shortly after the trauma appears to be a strong predictor of who will later develop PTSD (Brewin et al., 1999). Although SSRIs are commonly administered in general medical practice and have been demonstrated effective for the treatment of PTSD, there has not been systematic study of their use for the treatment of ASD, ASD symptoms, or the prevention of PTSD, and this study represents one of the first attempts to systematically evaluate their use for this indication.

Sixty study participants (for 30 randomized) will be drawn from patients admitted to the Massachusetts General Hospital medical/surgical inpatient units for a traumatic injury that occurred in the prior 3 weeks. Study participants must meet criteria for the A1, A2 and at least one additional category of Acute Stress Disorder symptoms (i.e., B, C and or D criteria), as determined by the Acute Stress Disorder Interview upon initial evaluation, to qualify for randomization in a 12 week, double-blind flexible-dose treatment trial of escitalopram (10-40 mg/d) versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients at least 18 years of age with a primary (the condition that is most central to the patient's current distress) symptoms of Acute Stress Disorder as defined by DSM-IV criteria: A1, A2 and at least one additional category of Acute Stress Disorder symptoms (i.e., B, C and or D criteria).
* Patients must have had a medical trauma (even if fully resolved or minor) within the prior 3 weeks resulting in admission to the emergency room and/or inpatient hospital as part of their acute trauma resulting in ASD symptoms.

Exclusion Criteria:

* Patients will be excluded from entry into the study for current serious medical instability such as hemodynamic compromise, or serious head injury resulting in impaired mental status. Patients with a history of medical instability associated with their traumatic injury will be allowed study entry once the problem has resolved (as long as resolves within 3 weeks of trauma as per inclusion criteria).
* Patients with a trauma resulting in head injury related seizures, or with epilepsy (except a prior history of febrile seizures of infancy which are not exclusionary).
* Pregnant or lactating women or those of childbearing potential not using medically accepted forms of contraception will be excluded.
* Concurrent use of other antidepressants, with the exception of trazodone < 100mg/day for sleep, or amitriptyline in doses ≤ 50 mg daily for pain. Patients may remain on concomitant benzodiazepines (<2 mg/d clonazepam or its equivalent), or sleep aids (i.e., trazodone, zolpidem (Ambien), zaleplon (Sonata)) as long as the drug therapy was initiated at 1 week prior to randomization; the dose will be held constant through the study, and will be controlled for in the analysis.
* Lifetime diagnosis of schizophrenia or any other psychosis, mental retardation, organic mental disorders, bipolar disorder; obsessive-compulsive disorder, eating disorders, cutting or other significant self-injurious behavior, or alcohol/substance abuse disorders within the last 3 months are study exclusions. Patients with a current primary diagnosis of major depression, dysthymia, social anxiety disorder, panic disorder, and generalized anxiety disorder are excluded; thus, the presence of these disorders is permissible as long as the ASD symptoms constitute the predominant symptomatology.
* Patients with a history of hypersensitivity or prior poor response to escitalopram are excluded.
* Concurrent dynamic or supportive psychotherapy is permitted as long as it has been ongoing for at least 1 month prior to onset of study entry.
* Patients with a positive toxicology screen at baseline consistent with evidence of current substance abuse or dependence as determined by clinical interview.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2005-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of Acute Stress Disorder
Symptoms of Posttraumatic Stress Disorder

SECONDARY OUTCOMES:
Clinical Global Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- See also: Official Website for the Center for Anxiety and Traumatic Stress Disorders — http://www.mghanxiety.org